CLINICAL TRIAL: NCT00063323
Title: Maintenance Treatment for Prevention of Smoking Relapse
Brief Title: Maintenance Treatment for Abstinent Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Lirio S. Covey, Research Foundation for Mental Hygiene
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-13490-1; R01DA013490 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2003-06-25; First posted 2003-07-01 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Tobacco Use Disorder
Keywords: Maintenance treatment; Smoking relapse; Bupropion; Nicotine replacement
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bupropion (Active Comparator): Bupropion (brand name Zyban Sustained Release). Participants used bupropion SR 150 mg twice daily during the 16-week maintenance treatment.
  Interventions: Drug: Bupropion
- Nicotine gum (Active Comparator): Nicotine gum (brand name Nicorette) During the maintenance 16-week maintenance treatment phase, participants assigned to this arm received 2 mg. nicotine gum.
  Interventions: Drug: Bupropion
- Bupropion+Nicotine Gum (Active Comparator): Combined active treatments: Bupropion (Zyban SR) and nicotine gum (Nicorette). Participants were instructed to use the 150 mg bupropion pill twice daily and the 2 mg. gum as needed during the 16-week maintenance treatment phase.
  Interventions: Drug: Bupropion
- Double placebo (Placebo Comparator): Placebo gum + placebo pill. Identical placebo pill was used twice daily and identical placebo gum was used as needed.
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion

SUMMARY:
The purpose of this study is to determine the efficacy and cost-effectiveness of long-term pharmacotherapy (using Zyban and/or nicotine replacement) for reducing the relapse rate associated with stopping smoking.

DETAILED DESCRIPTION:
The goal of this study was to assess relapse prevention outcomes among individuals able to stop smoking when pharmacotherapy is extended beyond the standard duration of treatment. We hypothesized that maintenance treatment with prolonged bupropion use and/or "as needed" use of nicotine gum will reduce relapse to smoking. Participants were recruited through advertisements on radio, television, newspapers, the Internet, and various community outlets. Respondents were pre-screened by telephone using a standard interview. The first participant entered the OLT phase in February 2001; the final NTFU visit took place in October 2005.

The study was multi-phased consisting of: 1) eight-week open-label treatment (OLT) with bupropion and nicotine patch; 2) randomized double-blind assignment of OLT successes to 16 weeks of placebo-controlled maintenance treatment (MT); and 3) 24 weeks of non-treatment follow-up (NTFU). Participants received $25 compensation for completing the NTFU visits at Weeks 36 and 48. The Institutional Review Board of the New York State Psychiatric Institute approved the study. The study was performed at the Columbia University Medical Center Smoking Cessation Clinic in New York City.

ELIGIBILITY:
Inclusion Criteria:

* Patients who smoke at least 10 cigarettes daily and have attempted to quit smoking at least once

Exclusion Criteria:

* Seizure History
* Unstable Blood Pressure
* Current major depression
* Current alcohol/drug abuse or dependency
* Lifetime psychotic illness
* Current use of psychotropic drugs
* Unstable medical condition

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2000-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Survival abstinence rate with maintenance treatment | 48 weeks after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lirio S. S Covey, Ph.D., Principal Investigator — Research Foundation for Mental Hygiene, Inc.
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Result] Covey LS, Glassman AH, Jiang H, Fried J, Masmela J, LoDuca C, Petkova E, Rodriguez K. A randomized trial of bupropion and/or nicotine gum as maintenance treatment for preventing smoking relapse. Addiction. 2007 Aug;102(8):1292-302. doi: 10.1111/j.1360-0443.2007.01887.x. PMID 17624979
- [Result] Covey LS, Botello-Harbaum M, Glassman AH, Masmela J, LoDuca C, Salzman V, Fried J. Smokers' response to combination bupropion, nicotine patch, and counseling treatment by race/ethnicity. Ethn Dis. 2008 Winter;18(1):59-64. PMID 18447101
- [Result] Covey LS, Manubay J, Jiang H, Nortick M, Palumbo D. Smoking cessation and inattention or hyperactivity/impulsivity: a post hoc analysis. Nicotine Tob Res. 2008 Dec;10(12):1717-25. doi: 10.1080/14622200802443536. PMID 19023824
- [Result] Covey LS, Weissman J, LoDuca C, Duan N. A comparison of abstinence outcomes among gay/bisexual and heterosexual male smokers in an intensive, non-tailored smoking cessation study. Nicotine Tob Res. 2009 Nov;11(11):1374-7. doi: 10.1093/ntr/ntp137. Epub 2009 Sep 24. PMID 19778993
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961